CLINICAL TRIAL: NCT05683613
Title: Watering of the Eyes Following Uneventful Phacoemulsification Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Helmy Mahmoud, Resident doctor at ophthalmology department in sohag university hospital, Sohag University
Other Study IDs: AHMahmoud
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Watery Eyes
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study aiming to assess the incidence and possible causes of post phacoemulsification watery eye.

DETAILED DESCRIPTION:
This study will be conducted on patients who will undergo cataract extraction at Sohag university hospitals to evaluate the incidence of watery eyes in patients after phacoemulsification by one week , one month and three month.

* Study Design: observational study.
* Inclusion Criteria:

Patients with age-related cataract.

* Exclusion Criteria:

  1. patients with watering of eyes or ocular surface diseases or watering of the eyes .
  2. patients with previous ocular surgeries.
  3. patients with glaucoma, uveitis, corneal or retinal pathologies.
* Preoperative Evaluation:

Each patient will be subjected to the following:

Detailed history taking and full ophthalmological examination. Fluorescein dye disappearance test. Syringing and probing. Schirmer's test. Tear break up time test. Measurement of punctal diameter by AS-OCT.

* Operative procedures:

  1. regional anesthesia.
  2. phaco technique : stop and shop.
  3. cumulative dissipated energy (CDE ) &fluid flow.
* Follow-up regimen: will be as follows:

  1. patients will be examined after surgery on: 1st postoperative week, 1st month, 3rd month.
  2. The following will be recorded for each patient:

     1. symptoms of watery eyes, visual acuity, IOP, slit lamp examination.
     2. dye disappearance test.
     3. Schirmer's test.
     4. tear break up time test.
     5. anterior segment OCT.

ELIGIBILITY:
Inclusion Criteria:

* patients with age related cataract.

Exclusion Criteria:

* patients with watering of the eyes or ocular surface disease.

  * patients with previous ocular surgeries .
  * patients with glaucoma, uveitis, cornealor retinal pathologies.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50_ 80 year old Patients with age related cataract with no watery eyes subjected for phacoemulsification cataract surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence and possible causes of post phacoemulsification watery eye. | Five months
  Patients are examined preoperatively and postoperatively by flourescein disappearance test, probing and syringing, schirmer's test,tear breakup time test and anterior segment optical coherence tomography to detect incidence and causes of post phacoemulsification watery eye.